CLINICAL TRIAL: NCT06517524
Title: Effects of Low-pressure Pneumoperitoneum Associated With Deep Pipecuronium-induced Neuromuscular Blockade on Hemodynamic Parameters for High Cardiovascular Risk Patient Undergoing General Anesthesia
Status: Completed | Type: Observational
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, Head, Division of General, Vascular and Thoracic Anesthesia, University of Debrecen
Organization: University of Debrecen (Other)
Other Study IDs: AITT/2022/6; OGYEI/3968-1/2023 (Other: National Institute of Pharmacy and Nutrition); DE RKEB/IKEB:6252-2022 (Other: Regional and Institutional Ethics Committee University of Debrecen Clinical Center)
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Residual Neuromuscular Block; Cardiovascular Diseases; Neuromuscular Blockade Monitoring
Keywords: neuromuscular monitoring; deep neuromuscular blockade; laparoscopic surgery
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Deep neuromuscular block (DNMB) during laparoscopy induces less haemodynamic stress by facilitating low-pressure pneumoperitoneum. the investigators tested the feasibility of pipecuronium-induced deep (post-tetanic count ≥1, train-of-four count = 0) NMB to allow low intraabdominal pressures and maintain cardiovascular stability in patients with low cardiac ejection fraction.MethodsTen adult, NYHA 3-4 surgical patients requiring non-elective abdominal surgery, were included. Pipecuronium bromide (PIPE) 0.09 mg/kg was used for muscle relaxation and maintenance of DNMB. Top-up doses of PIPE were administered when the post-tetanic count was 4-8.

Intraabdominal pressures (IAP) were kept below 10 mmHg. Mean arterial pressure (MAP) was measured intra-arterially. Outcome measures used: weight in kilograms, height in meters, need for circulatory suppert (yes/no), success of maintenance (yes/no). Surgical field view was rated on a 5-point scale (1= extremely poor, 5 = optimal)

DETAILED DESCRIPTION:
Patients with a high cardiovascular risk who undergo lparoscopic cholecystectomy before cardiac surgery were included in the study. It is known from the literature that low pressure pneumoperitoneum has less circulatory effects than normal pressure pneumoperitoneum.The abdominal muscles are well relaxed by a deep neuromuscular block using a pypecuronium bromide muscle relaxant. The quality of the surgical field of view is expected to improve. With deep muscle relaxation, low-pressure pneumoperitoneum can be easily maintained, thus the investigators hypothesise that patients will remain haemodynamically stable during surgery.

Primary endpoint of the study

Maintenance of low-pressure (6-10 mmHg) pneumoperitoneum during surgery using deep NMB with pipecuronium as neuromuscular blocking agent.

Secondary endpoint of the study

Number of cases with successful reversal of deep neuromuscular block to TOFR ≥0.9 within 3 min after administration of 2 mg/kg sugammadex.

Additional endpoints

Changes in hemodynamic parameters during surgery, need for pharmacologic circulatory support. Quality of the surgical field of view rated by the surgeon.

ELIGIBILITY:
Inclusion Criteria:

* high cardiovascular risk, class III- IV, according to the New York Heart Association classification of heart failure
* Age: between 18- 65 years old.
* ASA (American Society of Anesthesia score) 1- 3
* BMI between 18.5- 25
* Laparoscopic surgical interventions
* Endotracheal intubation
* Patient in supine position on operating table with one arm abducted and accessible.

Exclusion Criteria:

* Patients with diseases affecting neuromuscular functions (myopathies, severe liver and kidney failure).
* Patients on medications affecting the neuromuscular function (magnesium,aminoglycosides).
* Difficult airway or anticipated difficult airway.
* pregnancy (a pregnancy test was performed for every female patient in childbearing age to rule out pregnancy);
* Breastfeeding
* Acute surgical indications
* Chronic Obstructive Pulmonary Disease (COPD)
* Glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Effects of low-pressure pneumoperitoneum associated with deep Pipercuronium-induced neuromuscular blockade on hemodynamic parameters for high cardiovascular risk patients undergoing general anesthesia
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Succes of maintenance low-pressure pneumoperitoneum (6-10 mmHg) during laparascopic surgery | During laporoscopic surgery
  Succes of maintenance of low-pressure (6-10 mmHg) pneumoperitoneum during surgery using deep NMB with pipecuronium as neuromuscular blocking agent (yes/no).
  Pneumoperitoneum pressure will be registered continously throughout the study. The threshold for low IAP is predefined. The maintenance of low IAP will be assessed off-line (yes/no) as well as the IAP values as absolute numbers will be analized. If the intra-abdominal pressure is within this range (6-10 mmHg), maintenance of low-pressure pneumoperitoneum is considered successful (yes). Otherwise, maintaining a low-pressure pneumoperitoneum will prove unsuccessful.

SECONDARY OUTCOMES:
Succes of reversal of deep neuromuscular block mg/kg sugammadex. required. | During laporoscopic surgery
  Succes of reversal of deep neuromuscular block to TOFR ≥0.9 within 3 min after administration of 2 mg/kg sugammadex (yes/no). Reversal is considered successful (yes) if the time from administration of sugammadex to TOFR0.9 is less than 3 minutes. If this time is more than 3 minutes, the reversal is considered unsuccessful (no).

OTHER OUTCOMES:
Changes in hemodynamic parameters during surgery | During laporoscopic surgery
  Changes in hemodynamic parameters during surgery: invasive arterial blood pressure measurement is used to measure the patient's systolic and diastolic blood pressure values (mmHg). Patients are considered haemodynamically stable if these values remain within 15% of baseline.
Changes in Heart rate (beat/min) during surgery | During laporoscopic surgery
  Changes in hemodynamic parameters during surgery. Patients are considered haemodynamically stable if these values remain within 15% of baseline.
The mean arterial pressure recorded (mmHg) | During laporoscopic surgery
  Patients are considered haemodynamically stable if these values remain within 15% of baseline.
Need for pharmacologic circulatory support | During laporoscopic surgery
  The need for catecholamine administration during surgery: yes or no
Quality of the surgical field of view | During laporoscopic surgery
  Quality of the surgical field of view rated by the surgeon. We use five- point scale according to Baete et. al. study from 2017.
  The operating surgeon can choose between 1 to 5 according to the quality of the surgical field, where 1= very bad, 2=bad, 3= acceptable, 4 =good, 5=optimal.
  We record the score chosen by the surgeon.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, Full professor, Doctor of HAS, Principal Investigator — Department of Anesthesiology and Intensive Care University of Debrecen
Locations (1):
- University of Debrecen, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] Neudecker J, Sauerland S, Neugebauer E, Bergamaschi R, Bonjer HJ, Cuschieri A, Fuchs KH, Jacobi Ch, Jansen FW, Koivusalo AM, Lacy A, McMahon MJ, Millat B, Schwenk W. The European Association for Endoscopic Surgery clinical practice guideline on the pneumoperitoneum for laparoscopic surgery. Surg Endosc. 2002 Jul;16(7):1121-43. doi: 10.1007/s00464-001-9166-7. Epub 2001 May 20. PMID 12015619
- [Background] Hypolito OH, Azevedo JL, de Lima Alvarenga Caldeira FM, de Azevedo OC, Miyahira SA, Miguel GP, Becker OM Jr, Machado AC, Nunes Filho GP, Azevedo GC. Creation of pneumoperitoneum: noninvasive monitoring of clinical effects of elevated intraperitoneal pressure for the insertion of the first trocar. Surg Endosc. 2010 Jul;24(7):1663-9. doi: 10.1007/s00464-009-0827-2. Epub 2009 Dec 25. PMID 20035347
- [Background] Eryilmaz HB, Memis D, Sezer A, Inal MT. The effects of different insufflation pressures on liver functions assessed with LiMON on patients undergoing laparoscopic cholecystectomy. ScientificWorldJournal. 2012;2012:172575. doi: 10.1100/2012/172575. Epub 2012 Apr 24. PMID 22619616
- [Background] Sarli L, Costi R, Sansebastiano G, Trivelli M, Roncoroni L. Prospective randomized trial of low-pressure pneumoperitoneum for reduction of shoulder-tip pain following laparoscopy. Br J Surg. 2000 Sep;87(9):1161-5. doi: 10.1046/j.1365-2168.2000.01507.x. PMID 10971421
- [Background] Esmat ME, Elsebae MM, Nasr MM, Elsebaie SB. Combined low pressure pneumoperitoneum and intraperitoneal infusion of normal saline for reducing shoulder tip pain following laparoscopic cholecystectomy. World J Surg. 2006 Nov;30(11):1969-73. doi: 10.1007/s00268-005-0752-z. PMID 17043939
- [Background] Madsen MV, Staehr-Rye AK, Claudius C, Gatke MR. Is deep neuromuscular blockade beneficial in laparoscopic surgery? Yes, probably. Acta Anaesthesiol Scand. 2016 Jul;60(6):710-6. doi: 10.1111/aas.12698. Epub 2016 Feb 10. PMID 26864853
- [Background] Blobner M, Frick CG, Stauble RB, Feussner H, Schaller SJ, Unterbuchner C, Lingg C, Geisler M, Fink H. Neuromuscular blockade improves surgical conditions (NISCO). Surg Endosc. 2015 Mar;29(3):627-36. doi: 10.1007/s00464-014-3711-7. Epub 2014 Aug 15. PMID 25125097
- [Background] Bruintjes MH, van Helden EV, Braat AE, Dahan A, Scheffer GJ, van Laarhoven CJ, Warle MC. Deep neuromuscular block to optimize surgical space conditions during laparoscopic surgery: a systematic review and meta-analysis. Br J Anaesth. 2017 Jun 1;118(6):834-842. doi: 10.1093/bja/aex116. PMID 28575335
- [Background] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Ozdemir-van Brunschot DMD, Braat AE, van der Jagt MFP, Scheffer GJ, Martini CH, Langenhuijsen JF, Dam RE, Huurman VA, Lam D, d'Ancona FC, Dahan A, Warle MC. Deep neuromuscular blockade improves surgical conditions during low-pressure pneumoperitoneum laparoscopic donor nephrectomy. Surg Endosc. 2018 Jan;32(1):245-251. doi: 10.1007/s00464-017-5670-2. Epub 2017 Jun 22. PMID 28643056
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Background] Torensma B, Martini CH, Boon M, Olofsen E, In 't Veld B, Liem RS, Knook MT, Swank DJ, Dahan A. Deep Neuromuscular Block Improves Surgical Conditions during Bariatric Surgery and Reduces Postoperative Pain: A Randomized Double Blind Controlled Trial. PLoS One. 2016 Dec 9;11(12):e0167907. doi: 10.1371/journal.pone.0167907. eCollection 2016. PMID 27936214
- [Background] Abrishami A, Ho J, Wong J, Yin L, Chung F. Sugammadex, a selective reversal medication for preventing postoperative residual neuromuscular blockade. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD007362. doi: 10.1002/14651858.CD007362.pub2. PMID 19821409
- [Background] Tassonyi E, Pongracz A, Nemes R, Asztalos L, Lengyel S, Fulesdi B. Reversal of Pipecuronium-Induced Moderate Neuromuscular Block with Sugammadex in the Presence of a Sevoflurane Anesthetic: A Randomized Trial. Anesth Analg. 2015 Aug;121(2):373-80. doi: 10.1213/ANE.0000000000000766. PMID 25923435
- [Background] Tassonyi E, Asztalos L, Szabo-Maak Z, Nemes R, Pongracz A, Lengyel S, Fulesdi B. Reversal of Deep Pipecuronium-Induced Neuromuscular Block With Moderate Versus Standard Dose of Sugammadex: A Randomized, Double-Blind, Noninferiority Trial. Anesth Analg. 2018 Dec;127(6):1344-1350. doi: 10.1213/ANE.0000000000003719. PMID 30169407
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Naguib M, Brull SJ, Kopman AF, Hunter JM, Fulesdi B, Arkes HR, Elstein A, Todd MM, Johnson KB. Consensus Statement on Perioperative Use of Neuromuscular Monitoring. Anesth Analg. 2018 Jul;127(1):71-80. doi: 10.1213/ANE.0000000000002670. PMID 29200077
- [Derived] Asztalos L, Szabo-Maak Z, Berhes M, Kanyari Z, Nagy G, Pongracz A, Nemes R, Brull SJ, Fulesdi B. Deep neuromuscular block with pipecuronium in patients undergoing laparoscopic surgery - A prospective case series. Anaesth Crit Care Pain Med. 2025 Apr;44(2):101493. doi: 10.1016/j.accpm.2025.101493. Epub 2025 Feb 19. PMID 39983904